CLINICAL TRIAL: NCT03825068
Title: Erector Spinae Plane Block in Minimal Invasive Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer of anaesthesia and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RRLL
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthetics, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP block group (Active Comparator): patients receive ESP Bock with local anaesthetics
  Interventions: Procedure: ESP Block
- control group (Placebo Comparator): general anaestesia
  Interventions: Drug: general anesthetic

INTERVENTIONS:
Procedure: ESP Block — 20 ml of lacal anaesthetics will be placed below the erector spinae muscle under ultrasound guide
  Arms: ESP block group
Drug: general anesthetic — patient receive general anaesthetic only
  Arms: control group

SUMMARY:
Studying the effect of erector spinae plane block in patients undergoing minimal invasive cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective valve replacement

Exclusion Criteria:

* chroic renal failure
* chronic liver failure

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
VAS | 48 hours
  PAIN SCORES OF PATIENTS

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt